CLINICAL TRIAL: NCT00053339
Title: Phase III Randomized Study of Trastuzumab (Herceptin) With or Without Tamoxifen in Women With Progressive, Stage IV, Estrogen or Progesterone Receptor- and HER2/Neu-Positive Breast Cancer
Brief Title: Trastuzumab With or Without Tamoxifen in Treating Women With Progressive Stage IV Breast Cancer
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was not activated.
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CALGB-49903; CDR0000269409 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Stage IV Breast Cancer; Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Tamoxifen; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- trastuzumab (Experimental): Patients receive trastuzumab (Herceptin) IV over 60-90 minutes on day 1.
  Treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months for 5 years.
  Interventions: Drug: trastuzumab
- trastuzumab + tamoxifen (Experimental): Patients receive trastuzumab V over 60-90 minutes on day 1 and oral tamoxifen once daily on days 1-21.
  In both arms, treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months for 5 years.
  Interventions: Drug: tamoxifen; Drug: trastuzumab

INTERVENTIONS:
Drug: tamoxifen
  Arms: trastuzumab + tamoxifen
Drug: trastuzumab

SUMMARY:
RATIONALE: Monoclonal antibodies such as trastuzumab can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Estrogen can stimulate the growth of breast cancer cells. Hormone therapy using tamoxifen may fight breast cancer by blocking the uptake of estrogen. Combining trastuzumab with tamoxifen may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of trastuzumab with or without trastuzumab in treating women who have invasive stage IV breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare time to progression in women with progressive, stage IV, estrogen or progesterone receptor- and HER2/neu-positive breast cancer treated with trastuzumab (Herceptin) with or without tamoxifen.
* Correlate response with type of measurement (immunohistochemistry or fluorescent in situ hybridization) of HER2/neu expression in patients treated with these regimens.
* Compare objective response rate (complete or partial response) in patients treated with these regimens.

OUTLINE: This is a randomized study. Patients are stratified according to prior adjuvant treatment (yes vs no), ECOG performance status (0-1 vs 2), and prior aromatase inhibitor treatment (yes vs no). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive trastuzumab (Herceptin) IV over 60-90 minutes on day 1.
* Arm II: Patients receive trastuzumab as in arm I and oral tamoxifen once daily on days 1-21.

In both arms, treatment repeats every 3 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 5 years.

PROJECTED ACCRUAL: A total of 280 patients (140 per treatment arm) will be accrued for this study within 28 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed invasive stage IV breast cancer
* Hormone receptor status:
* HER2/neu positive (3+ by immunohistochemical [IHC] assay or fluorescent in situ hybridization [FISH])
* Estrogen receptor or progesterone receptor positive
* Measurable or evaluable disease
* Must have disease progression within 6 months of initiation of tamoxifen (administered in the adjuvant or metastatic setting) or during aromatase inhibitor therapy

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Performance status

* ECOG 0-2

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* SGOT and SGPT no greater than 2.5 times ULN

Cardiovascular

* LVEF normal by MUGA

Other

* Not pregnant or nursing
* Fertile patients must use effective nonhormonal contraception during and for at least 2 months after study completion
* No other concurrent active malignancy except nonmelanoma skin cancer
* Patients who have completed prior therapy and are at less than 30% risk of relapse are not considered to have an active malignancy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior trastuzumab (Herceptin) in the adjuvant or metastatic setting

Chemotherapy

* No more than 1 prior chemotherapy regimen in the metastatic setting
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* No more than 1 prior hormonal therapy regimen for metastatic disease
* Prior aromatase inhibitor therapy administered in the first-line metastatic or adjuvant setting is allowed provided there is disease progression on tamoxifen
* No other concurrent hormonal therapy except the following:
* Steroids for adrenal failure
* Hormones for nondisease-related conditions (e.g., insulin for diabetes)
* Intermittent use of dexamethasone as an antiemetic
* Vaginal estrogen (or EstringÂ®) for vaginal dryness

Radiotherapy

* No concurrent palliative radiotherapy except whole brain irradiation for CNS disease

Other

* Concurrent bisphosphonates allowed
* No concurrent cardioprotective drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Time to progression | Up to 5 years

SECONDARY OUTCOMES:
response | Up to 5 years
response rate | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Joanne E. Mortimer, MD, Study Chair — Sentara Cancer Center